CLINICAL TRIAL: NCT03531710
Title: An Extension Study of a Phase IIa Study in Patients With Mild Alzheimer's Disease to Evaluate the Safety, Tolerability, Immunogenicity, and Efficacy of UBITh® AD Immunotherapeutic Vaccine (UB-311)
Brief Title: An Extension Study of V203-AD Study to Evaluate the Safety, Tolerability, Immunogenicity, and Efficacy of UB-311
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: United Neuroscience has decided to terminate V203-AD-EXT study based on a treatment assignment error
Sponsor: United Neuroscience Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V203-AD-EXT
Record Dates: First submitted 2018-04-06; First posted 2018-05-22 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3 boosters (Experimental): Subjects will receive 3 doses of UB-311 and 2 doses of placebo.
  Interventions: Biological: UB-311; Drug: Placebo
- 3 priming doses followed by 2 boosters (Experimental): Subjects will receive 5 doses of UB-311.
  Interventions: Biological: UB-311

INTERVENTIONS:
Biological: UB-311 — Intramuscular injection
Drug: Placebo — Intramuscular injection
  Arms: 3 boosters

SUMMARY:
To evaluate the long-term safety, tolerability and potential efficacy, patients who previously participated in V203-AD study (NCT02551809) will be eligible to participate in the extension study and will receive 3 or 5 doses of UB-311 within a 96-week treatment period followed by a 12-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in V203-AD trial without major safety concerns;
* Stable doses of permitted medications for 3 months before screening;
* With a caregiver;
* Other inclusion criteria apply

Exclusion Criteria:

* Clinically significant neurological disease other than Alzheimer's disease
* Major psychiatric disorder
* Severe systemic disease
* Serious adverse reactions to any vaccine
* Other exclusion criteria apply

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital (KS-CGMH), Kaohsiung City
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Veterans General Hospital (TVGH), Taipei
  - Linkou Chang Gung Memorial Hospital (LK-CGMH), Taoyuan District

REFERENCES:
- See also: Site-specific UBITh amyloid-beta vaccine for immunotherapy of Alzheimer's disease. — http://www.ncbi.nlm.nih.gov/pubmed/17287052?dopt=Abstract
- See also: UB-311, a novel UBITh® amyloid β peptide vaccine for mild Alzheimer's disease. — http://www.ncbi.nlm.nih.gov/pubmed/?term=UB-311

RESULTS

PARTICIPANT FLOW:
Groups:
- M7E1: Treatment Group Arm 1 from V203-AD (M7) received 1 dose of UB-311 and 2 doses of placebo in V203-AD-EXT (E1)
- M7E3: Treatment Group Arm 1 from V203-AD (M7) received 3 doses of UB-311 in V203-AD-EXT (E3)
- M5E1: Treatment Group Arm 2 from V203-AD (M5) received 1 dose of UB-311 and 2 doses of placebo in V203-AD-EXT (E1)
- M5E3: Treatment Group Arm 2 from V203-AD (M5) received 3 doses of UB-311 in V203-AD-EXT (E3)
- M0E1: Treatment Group Arm 3 from V203-AD (M0) received 1 dose of UB-311 and 2 doses of placebo in V203-AD-EXT (E1)
- M0E3: Treatment Group Arm 3 from V203-AD (M0) received 3 doses of UB-311 in V203-AD-EXT (E3)
Period: Overall Study
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
Started | 10 | 2 | 7 | 5 | 8 | 2
Completed | 8 | 2 | 7 | 5 | 8 | 2
Not Completed | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3 | Total
Number analyzed (Participants) | 10 | 2 | 7 | 5 | 8 | 2 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (5.81) | 83.0 (7.07) | 75.4 (7.74) | 71.6 (6.8) | 74.9 (8.31) | 70.5 (4.95) | 74.2 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 4 | 3 | 6 | 2 | 24
  Male | 1 | 2 | 3 | 2 | 2 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 2 | 7 | 5 | 8 | 2 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 10 | 2 | 7 | 5 | 8 | 2 | 34
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — MMSE Total Score Presented. The MMSE is a 30-point questionnaire used extensively in clinical and research settings to measure cognitive impairment and is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document a participant's response to treatment. The total score range is 0 - 30 and lower scores indicating greater impairment.
  units on a scale | 17.2 (7.05) | 24 (4.24) | 18.71 (5.74) | 16.4 (7.47) | 18.13 (5.92) | 20.5 (2.12) | 18.21 (6.13)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Adverse Event (AE)/Serious Adverse Event (SAE) [Safety and Tolerability]).
Description: Summary of Treatment Emergent Adverse Events (TEAEs), based on reported adverse events and other safety information including local tolerability at injection site, MRI, vital signs, physical examination, 12-lead ECG and laboratory tests.
Time Frame: Overall Study Duration/Early Termination, over an average study duration of 326 days
Measure: Count of Participants; unit: Participants
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
Number analyzed (Participants) | 10 | 2 | 7 | 5 | 8 | 2
Participants | 4 | 1 | 4 | 3 | 5 | 2

2. Primary Outcome: Change From Baseline and Through to the End of the Study in Anti-Aβ Antibody Titers [The Immunogenicity of UB-311]
Description: For the immunogenicity assessment of the investigational product, UB-311, the level of anti-Aβ antibodies in the serum samples will be measured by a validated enzyme immunoassay manufactured by United Biomedical, Inc. (UBI). The level of anti-Aβ antibodies is assessed at every visit throughout the study period.
Time Frame: Overall Study Duration/Early Termination, over an average study duration of 326 days
Measure: Geometric Mean (Standard Deviation); unit: Geometric Mean Ratio in log10
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
Number analyzed (Participants) | 10 | 2 | 7 | 5 | 8 | 2
Geometric Mean Ratio in log10 | 0.56 (0.72) | 0.11 (0.35) | 0.15 (0.35) | 0.49 (0.32) | 0.10 (0.24) | 0.80 (0.09)

3. Other Pre Specified Outcome: Change From Baseline and Through to the End of the Study in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog);
Description: The ADAS-Cog 13 contains 13 items, with a total scoring range of 0 - 85 and higher scores indicating greater dysfunction. ADAS-Cog scores were evaluated at V1 and V8/ET. The observed values and change from baseline for ADAS-Cog scores by treatment groups in the extension study are presented
Time Frame: Overall Study Duration/Early Termination, over an average study duration of 326 days
Population: If more than one of 13 items of ADAS-Cog were missing/not available, ADASCog-13 total score was set to missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
Number analyzed (Participants) | 8 | 2 | 6 | 5 | 8 | 2
score on a scale | 2.86 (4.811) | -0.50 (2.121) | 2.50 (4.324) | 5.67 (3.512) | 3.50 (3.564) | 1.00 (1.414)

4. Other Pre Specified Outcome: Change From Baseline and Through to the End of the Study in Mini-Mental State Exam (MMSE)
Description: The MMSE is a 30-point questionnaire. The total score range is 0 - 30 and lower scores indicating greater impairment. MMSE scores were evaluated at V1 and V8/ET. The observed values and change from baseline for MMSE scores by treatment groups in the extension study are presented
Time Frame: Overall Study Duration/Early Termination, over an average study duration of 326 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
Number analyzed (Participants) | 10 | 2 | 7 | 5 | 8 | 2
score on a scale | -1.80 (3.225) | -1.50 (2.121) | -0.57 (1.618) | -3.00 (4.183) | -4.38 (4.868) | -2.00 (2.828)

5. Other Pre Specified Outcome: Change From Baseline and Through to the End of the Study in Clinical Dementia Rating - Sum of Boxes (CDR-SB)
Description: The CDR-SB includes 6 domains (0 - 3 points/domain), with a total scoring range of 0 - 18 and higher scores indicate greater impartment. CDR-SB scores were evaluated at V1 and V8/ET. The observed values and change from baseline for CDR-SB scores by treatment groups in the extension study are presented
Time Frame: Overall Study Duration/Early Termination, over an average study duration of 326 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
Number analyzed (Participants) | 10 | 2 | 7 | 5 | 8 | 2
score on a scale | 1.50 (2.483) | 0.00 (0.000) | 0.64 (1.345) | 2.00 (3.082) | 3.69 (4.869) | 0.75 (1.061)

ADVERSE EVENTS:
Time Frame: Adverse events collected from ICF to Early Termination Visit, mean study duration was 326.2 days.
Arm/Group | M7E1 | M7E3 | M5E1 | M5E3 | M0E1 | M0E3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/7 | 0/5 | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/2 | 2/7 | 0/5 | 1/8 | 1/2
Other Adverse Events (participants affected / at risk) | 4/10 | 1/2 | 2/7 | 3/5 | 5/8 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M7E1 (N=10) | M7E3 (N=2) | M5E1 (N=7) | M5E3 (N=5) | M0E1 (N=8) | M0E3 (N=2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M7E1 (N=10) | M7E3 (N=2) | M5E1 (N=7) | M5E3 (N=5) | M0E1 (N=8) | M0E3 (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura nonthrombocytopenic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Due to the incorrect treatment assignment and study early termination, this study was underpowered for analysis with secondary endpoints. Therefore, all secondary endpoints (change in ADAS-Cog, MMSE, CDR-SB) were considered as exploratory efficacy endpoints. 2. qEEG, cortical thickness, computerized cognitive tests, and the change of amyloid deposition with substantial amount of missing data/visit so they were omitted from group comparison analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site PIs must jointly publish results, unless permission is granted by Sponsor. If a joint publication is not done within 12 months after trial completion and database lock, then the site may publish its own results; provided that, a) Sponsor has 45 business days to review the proposed publication; b) the PI must delete any confidential information identified by Sponsor; and c) the PI must delay disclosure for 1 year if a patent application is filed by Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT03531710/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT03531710/SAP_001.pdf